CLINICAL TRIAL: NCT00800332
Title: Double-blind, Placebo-controlled Dose-finding Study With CYT003-QbG10 in Adult Patients With Rhinoconjunctivitis Due to House Dust Mite Allergy
Brief Title: Dose Finding Study With CYT003-QbG10 in Patients With House Dust Mite Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Clinical Development, Cytos Biotechnology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT003-QbG10 09
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Rhinoconjunctivitis; Allergies
Keywords: Rhinoconjunctivitis due to house dust mite allergy
MeSH Terms: conditions — Hypersensitivity | interventions — CYT003-QbG10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: CYT003-QbG10
- 2 (Experimental)
  Interventions: Drug: CYT003-QbG10
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CYT003-QbG10 — subcutaneous injection
  Arms: 1; 2
Drug: Placebo — subcutaneous injection
  Arms: 3

SUMMARY:
The purpose of the study is to test whether vaccinations with CYT003-QbG10 can improve allergy symptoms in patients with house dust mite allergy. The active treatment will be compared against placebo.

ELIGIBILITY:
Inclusion Criteria:

* Perennial allergic rhinoconjunctivitis due to clinically relevant allergy towards house dust mite allergens
* Further criteria as defined in the study protocol

Exclusion Criteria:

* Clinically manifested seasonal allergy/-ies which is/are expected to interfere with the patient's study treatment schedule and/or assessments
* Clinically relevant perennial allergy/-ies other than house dust mites allergy
* Contraindication to any study test or procedure
* Further criteria as defined in the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Rhinoconjunctivitis symptom and medication scores | Pre- / Post-Treatment

CONTACTS AND LOCATIONS:
Locations (8):
- Cytos Investigator Sites, Paide, Tartu, Tallin, Rakvere, Estonia
- Germany (2):
  - Cytos Investigator Sites, Fulda, Dresden, Ulm, Rodgau, Kassel, Eisenach
  - Cytos Investigator Sites, Wiesbaden, Frankfurt/M, Leipzig, Jena, Hamburg, Dulmen
- Cytos Investigator Sites, N. Faliro, Hiraklion, Athens, Greece
- Cytos Investigator Sites, Riga, Rezekne, Latvia
- Cytos Investigator Sites, Vilnius, Kaunas, Klaipeda, Lithuania
- Romania (2):
  - Cytos Investigator Sites, Galati, Cluj Napoca, Bahia Mare, Brasov, Piesti
  - Cytos Investigator Sites, Targu Mures, Bukarest, Craiova, Iasi

REFERENCES:
- [Derived] Klimek L, Willers J, Hammann-Haenni A, Pfaar O, Stocker H, Mueller P, Renner WA, Bachmann MF. Assessment of clinical efficacy of CYT003-QbG10 in patients with allergic rhinoconjunctivitis: a phase IIb study. Clin Exp Allergy. 2011 Sep;41(9):1305-12. doi: 10.1111/j.1365-2222.2011.03783.x. Epub 2011 Jun 14. PMID 21672053